CLINICAL TRIAL: NCT02733159
Title: A Phase II Trial of Pembrolizumab in Patients With Non-small Cell Lung Cancer and a Performance Status of 2
Brief Title: Pembrolizumab in Patients With Non-Small Cell Lung Cancer and a Performance Status 2
Acronym: PePS2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG_14-172; 2015-002241-55 (EudraCT Number); ISRCTN10047797 (Registry Identifier: ISRCTN Registry)
Record Dates: First submitted 2016-03-01; First posted 2016-04-11 (Estimated); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Performance Status 2; Pembrolizumab; MK-3475
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab (Experimental): Pembrolizumab: 200 mg Q3W, intravenous administration for a maximum of 2 years, or until progression or unacceptable toxicity.
  Interventions: Drug: pembrolizumab

INTERVENTIONS:
Drug: pembrolizumab — anti PD-1
  Other Names: MK-3475

SUMMARY:
This study is to determine that pembrolizumab is safe and tolerable at the selected dose for the treatment of Non-Small Cell Lung Cancer (NSCLC) in patients with a performance status of 2. All patients will receive pembrolizumab.

DETAILED DESCRIPTION:
Non-small cell lung cancer (NSCLC) is the most common type of lung cancer. There are several studies which demonstrate a role for the immune system in fighting lung cancer. However, there are multiple mechanisms by which cancer dampens this response. The PD-1 receptor-ligand interaction is one of the major pathways hijacked by tumours to help evade detection and elimination by the cells of the immune system. A number of compounds which block this pathway, including the drug pembrolizumab, have shown impressive results in some patients.

At present all of the trials with pembrolizumab reported thus far have been in patients with a good Performance Status (PS) of 0-1, a measure of daily activity. Unfortunately many patients with lung cancer have impaired performance status, making them ineligible for trials of new therapies including anti PD-1. Clinical trials of standard-of-care therapy have been successfully performed in the PS=2 only population demonstrating the feasibility of performing clinical trials in this population.

In this trial, the investigators would like to determine whether this drug can be used to treat Performance status 2 patients with a lower general daily activity. The purpose of this trial is to determine that pembrolizumab is safe and tolerable. The investigators would also like to see how well the treatment works, find out more information about tumour shrinkage, and learn more about the disease and how it changes over time.

ELIGIBILITY:
Core Inclusion Criteria:

* Histologically confirmed PD-L1 status defined NSCLC. Biopsy must be within 70 days of first treatment with pembrolizumab.
* Eastern Cooperative Oncology Group (ECOG) performance status 2.
* Life expectancy > 12 weeks.
* Uni-dimensionally measurable disease according to Response Evaluation Criteria in Solid Tumours (RECIST) v1.1
* Computerised Tomography (CT) scan of chest and abdomen within 28 days of starting pembrolizumab.
* Adequate haematological function:

  * Platelet count ≥100 x 109 /L.
  * Neutrophils ≥1.5 x 109/L.
  * Haemoglobin ≥ 90 g/L.
* Adequate hepatic function:

  * Serum bilirubin ≤1.5 x upper limit of normal (ULN).
  * Serum transaminases ≤2.5 x ULN.
* Adequate renal function: Creatinine clearance <1.5 times ULN concurrent with creatinine clearance >50 ml/min.
* Provision of signed and dated, written informed consent prior to any trial specific procedures, sampling and analyses.

Core Exclusion Criteria:

* Patients who do not meet the criteria of performance status = 2 on the ECOG Performance scale.
* Untreated symptomatic brain or leptomeningeal metastatic disease.
* Medical or psychiatric conditions compromising informed consent.
* Any medical condition which in the opinion of the investigator would compromise the ability of the patient to participate in the trial or which would jeopardise compliance with the protocol.
* Radiotherapy within 28 days of trial treatment.
* Active autoimmune disease that has required systemic treatment in past 2 years
* Chronic usage of steroids or other immunosuppressant medication.
* Previous history of pneumonitis.
* Any evidence of clinical autoimmunity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2024-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Middleton, Professor, Principal Investigator — University of Birmingham
Locations (10):
- United Kingdom (10):
  - The Christie NHS Foundation Trust, Manchester, Greater Manchester
  - Southampton University Hospitals NHS Trust, Southampton, Hampshire
  - Maidstone and Tunbridge Wells NHS Trust, Maidstone, Kent
  - University Hospital Birmingham NHS Foundation Trust, Birmingham, West Midlands
  - Velindre Cancer Centre, Cardiff
  - Western General Hospital, Edinburgh
  - United Lincolnshire Hospitals NHS Trust, Lincoln
  - Barts Health NHS Trust, London
  - University College London Hospitals, London
  - The Royal Marsden Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analysed during the current study are available from the corresponding author on reasonable request. The Cancer Research UK Clinical Trials Unit (CRCTU) is committed to responsible and controlled sharing of anonymised clinical trial data with the wider research community to maximise potential patient benefit while protecting the privacy and confidentiality of trial participants. Data anonymised in compliance with the Information Commissioners Office requirements, using a procedure based on guidelines from the Medical Research Council (MRC) Methodology Hubs, will be available for sharing with researchers outside of the trials team within 6 months of the primary publication. More detailed information on the CRCTU's Data Sharing Policy and the mechanism for obtaining data can be found on the CRCTU website: https://www.birmingham.ac.uk/research/activity/mds/trials/crctu/index.aspx.
Time Frame: Data will be available within 6 months of the primary publication.
Access Criteria: See Plan Description above.

REFERENCES:
- [Result] Middleton G, Brock K, Savage J, Mant R, Summers Y, Connibear J, Shah R, Ottensmeier C, Shaw P, Lee SM, Popat S, Barrie C, Barone G, Billingham L. Pembrolizumab in patients with non-small-cell lung cancer of performance status 2 (PePS2): a single arm, phase 2 trial. Lancet Respir Med. 2020 Sep;8(9):895-904. doi: 10.1016/S2213-2600(20)30033-3. Epub 2020 Mar 19. PMID 32199466
- See also: Pembrolizumab in performance status 2 patients with non-small cell lung cancer (NSCLC): Results of the PePS2 trial — https://doi.org/10.1093/annonc/mdy292.007
- Available data/document: Trial Website — https://www.birmingham.ac.uk/research/crctu/trials/PePS2/index.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial opened to recruitment on 7th November 2016 and the first patient was recruited on 4th January 2017. The trial was opened to recruitment at 10 National Health Service (NHS) hospitals across the United Kingdom. The last patient was recruited on 13th February 2018.
Groups:
- Pembrolizumab: Pembrolizumab: 200 mg Q3W (once every 3 weeks), intravenous administration for a maximum of 2 years, or until progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Pembrolizumab
Started | 62 (62 patients were registered to the trial.)
Completed | 60 (60/62 patients were considered the Analysis Population, 2 patients were excluded as they did not start trial treatment (listed as Not Completed in these results); 1 due to Adverse Event and 1 due to Lack of disease progression.)
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Lack of disease progression | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 62
Age, Continuous [Mean (Full Range); unit: years]
  Age at Registration (years) | 69.85 [43 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 34
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Histology [Count of Participants; unit: Participants]
  Adenocarcinoma | 43
  Adenosquamous Carcinoma | 0
  Squamous Cell Carcinoma | 12
  Not Otherwise Specified | 1
  Other | 6
Smoking Status [Count of Participants; unit: Participants]
  Current smoker | 11
  Ex-smoker | 45
  Never smoked | 3
  Not Known | 3
Smoking Pack Years [Mean (Full Range); unit: years] — Population: Only given for patients who self-identified as either current or ex-smokers.
  years
    number analyzed (Participants) | 56
    (all) | 43.78 [5 to 99]
Duration of Abstinence [Mean (Full Range); unit: years] — Population: Only given for patients who self-identified as ex-smokers
  years
    number analyzed (Participants) | 45
    (all) | 15.38 [0 to 65]
Charlson Co-Morbidity Index Score [Mean (Full Range); unit: units on a scale] — The Charlson Index (Charlson M.E. et al. doi:10.1016/0021-9681(87)90171-8) was used for the assessment of co-morbidities by the treating clinician of each patient; each co-morbidity is scored as 1, 2, 3 or 6 based on severity (higher score means greater severity). The sum is then calculated for each patient with co-morbidities, with a score of 1 added to the total score for each decade >40 years of age. Higher scores represent greater co-morbidities (worse outcome). A score of 0 means the patient had no co-morbidities. This validated and published index is detailed in the protocol Appendix 4.
  units on a scale | 7.58 [0 to 12]
Charlson Co-Morbidity Index Score [Count of Participants; unit: Participants] — The Charlson Index (Charlson M.E. et al. doi:10.1016/0021-9681(87)90171-8) was used for the assessment of co-morbidities by the treating clinician of each patient; each co-morbidity is scored as 1, 2, 3 or 6 based on severity (higher score means greater severity). The sum is then calculated for each patient with co-morbidities, with a score of 1 added to the total score for each decade >40 years of age. Higher scores represent greater co-morbidities (worse outcome). A score of 0 means the patient had no co-morbidities. This validated and published index is detailed in the protocol Appendix 4.
  Participants
    0 | 3
    1 | 0
    2 | 1
    3 | 4
    4 | 4
    5 | 4
    6 | 2
    7 | 3
    8 | 7
    9 | 19
    10 | 9
    11 | 2
    12 | 4
Sample Type [Count of Participants; unit: Participants] — Population: Only given for patients who had a successful PD-L1 staining of the tumour sample.
  Participants
    number analyzed (Participants) | 59
    Archived biopsy sample | 52
    New biopsy sample | 7
Percentage of Tumour Cells Expressing PD-L1 [Mean (Full Range); unit: %] — This trial was an all-comers design with PD-L1 expression measured and included as an integral part of the trial design at trial entry, as this was a potentially predictive biomarker for response with the trial drug. It is included in the eligibility criteria and is collected at baseline so is therefore it is listed as a baseline characteristic as it is crucial in the interpretation of the results. Population: Only given for patients who had a successful PD-L1 staining of the tumour sample.
  %
    number analyzed (Participants) | 59
    (all) | 24.89 [0 to 100]
PD-L1 Staining Result [Count of Participants; unit: Participants] — This trial was an all-comers design with PD-L1 expression measured and included as an integral part of the trial design at trial entry, as this was a potentially predictive biomarker for response with the trial drug. It is included in the eligibility criteria and is collected at baseline so is therefore it is listed as a baseline characteristic as it is crucial in the interpretation of the results. Population: Only given for patients who had a successful PD-L1 staining of the tumour sample.
  Participants
    number analyzed (Participants) | 59
    Negative (<1%) | 28
    Positive (1-49%) | 16
    Strong Positive (50-100%) | 15
Line of Therapy [Count of Participants; unit: Participants]
  First | 25
  Subsequent | 37
Previous Therapy [Number; unit: participants] — Population: Items are non-exclusive; a patient could have multiple previous therapies.
  participants
    Biological | 2
    Chemotherapy | 44
    Immunological | 1
    Radiotherapy | 28
    Surgery | 13

OUTCOME MEASURES:

1. Primary Outcome: Toxicity Rate
Description: Adverse events will be recorded in relation to each cycle of treatment and graded according to CTCAE criteria. The toxicity co-primary outcome measure for the trial is defined as the occurrence of a treatment-related dose delay or treatment discontinuation due to toxicity.
Time Frame: Date of patient registration until 6 months after the administration of the last treatment (a maximum of 2 years treatment and 6 months followup after end of treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 60
Participants
  Patients Experiencing Toxicity Event | 18
  Patients Not Experiencing Toxicity Event | 42

2. Primary Outcome: Durable Clinical Benefit
Description: Patients will have CT scans every 9 weeks from baseline until disease progression. On each occasion, overall tumour burden will be assessed using RECIST version 1.1. The efficacy co-primary outcome measure for the trial is durable clinical benefit defined as the occurrence of CR, PR or SD without prior progressive disease at or after the second scheduled CT scan (scheduled to occur at 18 weeks).
Time Frame: ≥18 weeks, up to maximum of 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 60
Participants
  Patients Experiencing Durable Clinical Benefits Event | 22
  Patients Not Experiencing DCB Event | 38

3. Secondary Outcome: Objective Response
Description: Objective response (OR) is the occurrence of Complete Response (CR) or Partial Response (PR) as the best overall response. OR will be based on responses confirmed using the subsequent 9-weekly scan but OR based on unconfirmed responses will also be reported.
Time Frame: ≥18 weeks, up to maximum of 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 60
Participants
  No | 44
  Yes | 16

4. Secondary Outcome: Health Related Quality of Life
Description: This is defined as the functional effect of a medical condition and/or its consequent treatment upon a patient. The purpose of Health Related Quality of Life (HRQoL) measurement is to quantify the degree to which the medical condition or its treatment impacts the individual's life in a valid and reproducible way. HRQoL will be assessed over time using Functional Assessment of Cancer Therapy - Lung (FACT-L) questionnaire and EQ-5D questionnaire.
Time Frame: Through study completion, up to a maximum of 2 years
Reporting Status: Not Posted

5. Secondary Outcome: Time to Progression
Description: This is defined as the time from commencement of trial treatment to the date of CT scan when progressive disease first recorded. Patients with no recorded progression at the time of analysis or who die without recorded progression will be censored at the date of the CT scan when they were last recorded with an evaluable measure that was not progression.
Time Frame: Time to progression up to 2 years
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 60
months | 11.9 [4.13 to 27.8]

6. Secondary Outcome: Progression-free Survival Time
Description: This is defined as the time from commencement of trial treatment to the date of CT scan when progressive disease first recorded or date of death without previously recorded progression. Patients who are alive with no recorded progression at the time of analysis will be censored at the date of the CT scan when they were last recorded with an evaluable measure that was not progression.
Time Frame: Progression-free survival time up to 2 years
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 60
months | 4.39 [3.48 to 9.9]

7. Secondary Outcome: Overall Survival Time
Description: This is defined as the time from commencement of trial treatment to the date of death. Patients who are alive at the time of analysis will be censored at the date last seen alive.
Time Frame: Survival time up to 2 years or date of death
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 60
months | 9.8 [6.77 to 13]

8. Secondary Outcome: Duration of Objective Response
Description: This is defined as the time from commencement of trial treatment to the date of the subsequent CT scan when progressive disease is first confirmed or date of death without previously recorded progression. This outcome is calculated and reported separately for patients who achieve an Objective Response (OR) or Stable Disease (SD). Patients experiencing OR or SD who are alive with no recorded progression at the time of analysis will be censored at the date of the CT scan when they were last recorded with an evaluable measure that was not progression.
Time Frame: Survival time up to 2 years or date of death
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 60
months | 14.6 [12.1 to NA] — The upper estimate of the confidence interval was not attained as there was an insufficient number of participants with events

9. Secondary Outcome: Duration of Stable Disease
Description: as for outcome 8
Time Frame: Survival time up to 2 years or date of death
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 60
months | 4.39 [3.97 to 6.77]

ADVERSE EVENTS:
Time Frame: Date of patient registration until 6 months after the administration of the last treatment (a maximum of 2 years treatment and 6 months followup after end of treatment)
Description: All medical occurrences which met the Adverse Event (AE) definition were reported including abnormal laboratory findings deemed clinically significant by Investigators (abnormal laboratory findings not clinically significant are not AEs) or any pre-existing AEs that worsened by at least 1 CTCAE grade from baseline. SAE expectedness was decided independently using the Reference Safety Information. 2/62 patients were excluded from the Analysis Population as they did not commence trial treatment.
Arm/Group | Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 48/60
Serious Adverse Events (participants affected / at risk) | 51/60
Other Adverse Events (participants affected / at risk) | 58/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=60)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (15)
Other - Death (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (5)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Other - Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Fever (General disorders) | 3 (3)
Lung infection (Infections and infestations) | 3 (3)
Confusion (Psychiatric disorders) | 1 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Stroke (Nervous system disorders) | 1 (2)
Vestibular disorder (Ear and labyrinth disorders) | 1 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Other - Death (Cardiac disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysphasia (Nervous system disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Other - Hepatobiliary disorders (Hepatobiliary disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Other - Chest Infection (Infections and infestations) | 1 (1)
Other - Infection (Infections and infestations) | 1 (1)
Other - Pneumonia (Infections and infestations) | 1 (1)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Other - Malignant neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Other - Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Other - Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
(General disorders) | 7 (7) — Death was reportable as an SAE, however, some of the SAEs were submitted retrospectively in error and the cause of death was unknown.
Other - Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Other - Shortness of Breath (Infections and infestations) | 1 (1)
Other - Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other - Acute Kidney Injury (Gastrointestinal disorders) | 1 (1)
Other - Nervous System (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=60)
Other - Creatinine decreased (Blood and lymphatic system disorders) | 1 (1)
Other - Haemoptysis (Blood and lymphatic system disorders) | 1 (1)
Other - Hypercalcemia (Blood and lymphatic system disorders) | 1 (1)
Other - Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 5 (8)
Cardiac arrest (Cardiac disorders) | 1 (1)
Other - Ejection systolic murmor (Cardiac disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Other - Hearing reduction (Ear and labyrinth disorders) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1)
Other - Adrenal insufficiency (Endocrine disorders) | 1 (1)
Hypophysitis (Endocrine disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 2 (3)
Hypothyroidism (Endocrine disorders) | 8 (9)
Other - Age related reduced visual acuity (Eye disorders) | 1 (1)
Other - Thromboembolic event left eye (Eye disorders) | 1 (1)
Watering eyes (Eye disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Other - Altered taste (Gastrointestinal disorders) | 1 (1)
Other - Decreased appetite (Gastrointestinal disorders) | 1 (1)
Other - Gastric reflux (Gastrointestinal disorders) | 1 (1)
Other - Reflux (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (3)
Dyspepsia (Gastrointestinal disorders) | 2 (5)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 14 (21)
Vomiting (Gastrointestinal disorders) | 14 (20)
Constipation (Gastrointestinal disorders) | 15 (24)
Nausea (Gastrointestinal disorders) | 15 (21)
Chills (General disorders) | 1 (1)
Flu like symptoms (General disorders) | 1 (1)
Other - Abdominal pain (General disorders) | 1 (1)
Other - Chest wall discomfort (occasional) (General disorders) | 1 (1)
Other - Cough (General disorders) | 1 (1)
Other - Dehydration (General disorders) | 1 (1)
Other - Edema feet (General disorders) | 1 (1)
Other - Hair thinning (General disorders) | 1 (1)
Other - Head cold (General disorders) | 1 (1)
Other - Itch (General disorders) | 1 (1)
Other - Leg cramps (General disorders) | 1 (1)
Other - Poor appetite (General disorders) | 1 (1)
Other - Raised sputum viscosity (General disorders) | 1 (1)
Other - Sore throat (General disorders) | 1 (1)
Other - Swollen feet and ankles (General disorders) | 1 (1)
Other - Weight loss (General disorders) | 1 (1)
Infusion related reaction (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 3 (3)
Malaise (General disorders) | 5 (6)
Edema limbs (General disorders) | 7 (8)
Fever (General disorders) | 9 (11)
Pain (General disorders) | 9 (10)
Fatigue (General disorders) | 36 (62)
Other - Bilirubin increased (Hepatobiliary disorders) | 1 (1)
Other - Drug induced liver injury (Hepatobiliary disorders) | 1 (1)
Other - Raised alk phosphate (Hepatobiliary disorders) | 1 (1)
Other - Rash (Immune system disorders) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1)
Other - Chest infections (Infections and infestations) | 1 (1)
Other - Chest Sepsis (Infections and infestations) | 1 (1)
Other - Cystitis (Infections and infestations) | 1 (1)
Other - Genital candida (Infections and infestations) | 1 (1)
Other - Infected picc line (Infections and infestations) | 1 (1)
Other - Lower respiratory track infection (Infections and infestations) | 1 (2)
Other - Lower respiratory tract infection (Infections and infestations) | 1 (1)
Other - Oral candida (Infections and infestations) | 1 (1)
Other - Oral candidiasis (Infections and infestations) | 1 (1)
Other - Picc line infection (Infections and infestations) | 1 (1)
Other - Presumed uti (Infections and infestations) | 1 (1)
Other - Thrush (Infections and infestations) | 1 (1)
Other - Undefined infection (Infections and infestations) | 1 (1)
Other - Unwell (Infections and infestations) | 1 (1)
Other - Viral infection (Infections and infestations) | 1 (1)
Other - Viral infection around mouth (Infections and infestations) | 1 (1)
Papulopustular rash (Infections and infestations) | 1 (1)
Other - Oral thrush (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 3 (3)
Other - Chest infection (Infections and infestations) | 6 (11)
Upper respiratory infection (Infections and infestations) | 6 (7)
Lung infection (Infections and infestations) | 10 (12)
Urinary tract infection (Infections and infestations) | 10 (16)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (2)
Blood corticotrophin decreased (Investigations) | 1 (1)
GGT increased (Investigations) | 1 (1)
Other - Cortisol low (Investigations) | 1 (1)
Other - Hyperbilirubinemia (Investigations) | 1 (1)
Other - Ldh raised - 794 (uln 480) (Investigations) | 1 (1)
Other - Thyroid stimulating hormone increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Serum amylase increased (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Creatinine increased (Investigations) | 3 (4)
Weight loss (Investigations) | 3 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Other - Low b12 (Metabolism and nutrition disorders) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 6 (9)
Hyponatremia (Metabolism and nutrition disorders) | 6 (12)
Anorexia (Metabolism and nutrition disorders) | 20 (28)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Other - Bruising to left arm (garden gate hit it) (Musculoskeletal and connective tissue disorders) | 1 (1)
Other - Discitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Other - Generalised muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2)
Other - Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Other - Heavy and painful left calf (Musculoskeletal and connective tissue disorders) | 1 (1)
Other - Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Other - Left arm pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Other - Left hip/ pelvic pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Other - Left sided gluteal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Other - Leg ache (Musculoskeletal and connective tissue disorders) | 1 (1)
Other - Muscle pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Other - Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (2)
Other - Right hand weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (4)
Other - Knee pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Other - Left shoulder pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (25)
Other - Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Concentration impairment (Nervous system disorders) | 1 (1)
Dysphasia (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Other - Involuntary neck movements (Nervous system disorders) | 1 (1)
Other - Pins & needles in right arm during antibiotic infusion (Nervous system disorders) | 1 (1)
Other - Tingling in extremeties (Nervous system disorders) | 1 (1)
Nystagmus (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 2 (2)
Paresthesia (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 5 (6)
Dizziness (Nervous system disorders) | 6 (9)
Confusion (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 4 (4)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (3)
Other - Raised creatinine (Renal and urinary disorders) | 1 (1)
Other - Renal failure (Renal and urinary disorders) | 1 (1)
Other - Urinary infection (Renal and urinary disorders) | 1 (1)
Other - Worsening of renal function (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 4 (6)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other - Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other - Cap-community acquired pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other - Chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other - Exacerbation of copd (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other - Increased sputum-brown (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other - Lower respiratory track infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other - Lower respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other - Lung crackles (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other - Mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other - Reduced air entry and a few creps (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other - Reduced air entry to right lung (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other - Reduced air entry to the right lower lobe (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other - Reduced breath sounds left upper lobe (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other - Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other - Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other - Right basal chest infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other - Scattered creps (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other - Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other - Shortness of breath on minimal exertion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other - White phlegm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Other - Chest infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Other - Exacerbation of chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Other - Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Other - Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (31)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 29 (48)
Other - Abdominal rash (Skin and subcutaneous tissue disorders) | 1 (1)
Other - Blisters on hands (Skin and subcutaneous tissue disorders) | 1 (1)
Other - Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Other - Dry skin on legs (Skin and subcutaneous tissue disorders) | 1 (1)
Other - Dry skin under right eye (Skin and subcutaneous tissue disorders) | 1 (2)
Other - Fungal skin rash (Skin and subcutaneous tissue disorders) | 1 (1)
Other - Infected sebaceous cycst (Skin and subcutaneous tissue disorders) | 1 (1)
Other - Itch (Skin and subcutaneous tissue disorders) | 1 (1)
Other - Itch skin (Skin and subcutaneous tissue disorders) | 1 (1)
Other - Itching (Skin and subcutaneous tissue disorders) | 1 (1)
Other - Itchy face (Skin and subcutaneous tissue disorders) | 1 (1)
Other - Itchy skin (Skin and subcutaneous tissue disorders) | 1 (1)
Other - Papulopustular (Skin and subcutaneous tissue disorders) | 1 (1)
Other - Pitting oedema (Skin and subcutaneous tissue disorders) | 1 (1)
Other - Pressure ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Other - Psoriasis rash (Skin and subcutaneous tissue disorders) | 1 (1)
Other - Rash on legs (Skin and subcutaneous tissue disorders) | 1 (1)
Other - Rash on the legs and arms (Skin and subcutaneous tissue disorders) | 1 (1)
Other - Red legs and mild oedema (Skin and subcutaneous tissue disorders) | 1 (1)
Other - Skin lesion to scalp (Skin and subcutaneous tissue disorders) | 1 (1)
Other - Sore feet and toes (Skin and subcutaneous tissue disorders) | 1 (1)
Other - Sore naval (Skin and subcutaneous tissue disorders) | 1 (1)
Other - Ulcer on left foot (Skin and subcutaneous tissue disorders) | 1 (1)
Other - X2 sore spots to upper right chest (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (5)
Other - Skin rash (Skin and subcutaneous tissue disorders) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (5)
Other - Rash (Skin and subcutaneous tissue disorders) | 3 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (7)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 12 (14)
Hypertension (Vascular disorders) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 1 (2)
Vasculitis (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 3 (3)
Thromboembolic event (Vascular disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-07-10): https://cdn.clinicaltrials.gov/large-docs/59/NCT02733159/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/59/NCT02733159/SAP_001.pdf